CLINICAL TRIAL: NCT01469130
Title: A Phase I Study of Oral MEK162 in Japanese Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Array Biopharma, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Organization: Array BioPharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMEK162X1101
Record Dates: First submitted 2011-11-08; First posted 2011-11-10 (Estimated); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Advanced Solid Tumor
Keywords: MEK, Advanced solid tumor
MeSH Terms: interventions — binimetinib

ARMS (1):
- MEK162 (Experimental): MEK162 will be administered orally once on Day 1 of Cycle 1 and continuously on a BID schedule, starting on Day 2 of Cycle 1 and on Day 1 of subsequent cycles. Each cycle will be 28 days in duration. Dose will be escalated and starting dose is 30 mg. Any doses that are missed should be skipped and should not be replaced or made up during the evening dosing or on a subsequent day, whichever applies.
  The prescribed BID doses should be taken 12 ± 2 hrs apart.
  Interventions: Drug: MEK162

INTERVENTIONS:
Drug: MEK162 — MEK162 in an oral formulation. It is a film-coated capsule-shape tablets (i.e. caplets).

SUMMARY:
In this study, MEK162 will be administered to Japanese patients with advanced solid tumors whose disease has progressed despite standard therapy or for whom no standard therapy exists. The trial will investigate the safety and tolerability and determine the MTD of MEK162 in Japanese patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically-confirmed, advanced unresectable solid tumors who have progressed within three months before screening/baseline visit.
* Availability of a representative formalin fixed paraffin embedded tumor tissue sample.
* At least one measurable or non-measurable lesion
* Age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2
* Good organ (hepatic, kidney, BM) function at screening/baseline visit.

Exclusion Criteria:

* Brain metastasis unless treated and free of signs/symptoms attributable to brain metastasis in the absence of corticosteroid therapy and anti-epileptic therapy.
* Impaired cardiac function or clinically significant cardiac disease incl. unstable angina pectoris ≤ 3 months prior to starting study drug and Acute Myocardial Infarction (AMI) ≤ 3 months prior to starting study drug.
* Women who are pregnant or breast feeding or adults of reproductive potential not employing an effective method of birth control.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-11; Primary Completion 2014-04 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Dose limiting toxicities | 4 weeks
  Incidence of frequency of Dose limiting toxicities during first 4 weeks will be measured according to the commen terminology criteria for adverse events (CTCAE).

SECONDARY OUTCOMES:
Incidence and severity of adverse events and serious adverse events, changes in laboratory values | 4 months
  Incidence and severity of adverse events and serious adverse events, changes in laboratory values will be measured during the treatment.
Plasma concentration of MEK162 and AR00426032active metabolite of MEK162 and derived PK parameters of MEK162 and the active metabolite. | 2 months
  Plasma concentration of MEK162 and active metabolite of MEK162 and derived PK parameters of MEK162 and the active metabolite will be measured with serial plasma samples during treatment for first 2 months.
Tumor responses according to RECIST 1.1 | 4 months
  Tumor responses will be measured according to RECIST 1.1
Levels of p-ERK in tumor and skin | 4 months
  Levels of p-ERK in tumor during treatment and skin for first 2 weeks will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- Japan (2):
  - Pfizer Investigative Site, Nagoya, Aichi-ken
  - Pfizer Investigative Site, Yufu, Oita Prefecture